CLINICAL TRIAL: NCT02499718
Title: Non-invasive Positive Pressure Ventilation for the Treatment of Severe Stable Chronic Obstructive Pulmonary Disease
Brief Title: Non-invasive Positive Pressure (NPPV ) for Severe Stable Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Southern Medical University, China (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Dongguan People's Hospital (Other Government)
Responsible Party: Principal Investigator, LuQian Zhou, Assistant Professor of Guangzhou Institute of Respiratory Disease, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRID-201506
Record Dates: First submitted 2015-06-09; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hypercapnic Respiratory Failure
Keywords: Chronic Obstructive Pulmonary Disease; Non-invasive positive pressure ventilation; quality of life; long-term oxygen therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Noninvasive ventilator (Experimental): noninvasive positive pressure ventilation combined with long-term oxygen therapy for severe stable chronic obstructive pulmonary disease
  Interventions: Device: BiPAP mode
- LTOT (No Intervention): long-term oxygen therapy for severe stable chronic obstructive pulmonary disease

INTERVENTIONS:
Device: BiPAP mode — Noninvasive ventilator
  Arms: Noninvasive ventilator

SUMMARY:
Assessment of the effect and safety of noninvasive positive pressure ventilation for severe stable chronic obstructive pulmonary disease

ELIGIBILITY:
Inclusion Criteria:

* clinically stable, hypercapnic GOLD stage IV COPD, aged 18 years or older, baseline arterial carbon dioxide pressure (PaCO2) of 6.7 kPa (50 mmHg) or higher and a pH higher than 7·35, measured after at least 1 h rest in a sitting position.

Exclusion Criteria:

* thorax or the lung other than COPD
* No smoking or Cigarette≤10/day
* obesity with a bodymass index (BMI) ≥40 kg/m²
* malignant co-morbidities,severe heart failure (New York Heart Association stage IV),unstable angina, and severe arrhythmias.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Severe Respiratory Insufficiency (SRI) Questionnaire | 1 year

SECONDARY OUTCOMES:
Blood gas analysis | 1 year
Pulmanory function | 1 year
Baseline Dyspnea Index/Transition Dyspnea Index | 1 year
Chromic Respiratory Questionnaire | 1 year
Chronic Obstructive Pulmonary Disease (COPD) Assessment Test | 1 year
6 Minute-Walking Distance and Borg Score | 1 year
The frequency of exacerbation | 1 year
The frequency of readmission | 1 year
The frequency of ICU readmission | 1 year
survival rate | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Chen R, Guan L, Wu W, Yang Z, Li X, Luo Q, Liang Z, Wang F, Guo B, Huo Y, Yang Y, Zhou L. The Chinese version of the Severe Respiratory Insufficiency questionnaire for patients with chronic hypercapnic chronic obstructive pulmonary disease receiving non-invasive positive pressure ventilation. BMJ Open. 2017 Aug 28;7(8):e017712. doi: 10.1136/bmjopen-2017-017712. PMID 28851800
- [Derived] Zhou L, Li X, Guan L, Chen J, Guo B, Wu W, Huo Y, Zhou Z, Liang Z, Zhou Y, Tan J, Chen X, Song Y, Chen R. Home noninvasive positive pressure ventilation with built-in software in stable hypercapnic COPD: a short-term prospective, multicenter, randomized, controlled trial. Int J Chron Obstruct Pulmon Dis. 2017 Apr 27;12:1279-1286. doi: 10.2147/COPD.S127540. eCollection 2017. PMID 28490871